CLINICAL TRIAL: NCT00343122
Title: Evaluation of Two Methods for the Echocardiographic Assessment of Intrapulmonary Vasodilatation in Patients With Liver Cirrhosis: Agitated Saline Versus Polygelatine
Brief Title: Echocardiographic Assessment of Intrapulmonary Vasodilatation: Agitated Saline Versus Polygeline
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Other Study IDs: EK 4462005
Record Dates: First submitted 2006-06-20; First posted 2006-06-22 (Estimated); Last update posted 2007-09-17 (Estimated); Status verified 2007-09

CONDITIONS: Liver; Cirrhosis
Keywords: liver; cirrhosis; hepatopulmonary syndrome
MeSH Terms: conditions — Fibrosis; Hepatopulmonary Syndrome

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

INTERVENTIONS:
Procedure: echocardiography for intrapulmonary vasodilatation

SUMMARY:
The purpose of the study is to evaluate agitated saline versus polygeline for detection of intrapulmonary vasodilatation in patients with cirrhosis.

DETAILED DESCRIPTION:
Intrapulmonary vasodilatation is a frequent finding in patients with cirrhosis. Its diagnosis is established via contrast enhanced echocardiography. One used method is the contrast agent agitated saline and another frequently used method is the contrast agent polygeline. The purpose of this study is to compare these two echocardiographic contrast agents with respect to their ability to detect intrapulmonary vasodilatation.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* presence of liver cirrhosis
* evaluation for liver transplantation or transjugular intrahepatic portosystemic shunt

Exclusion Criteria:

* inadequate echocardiographic image quality
* allergies to echocardiographic contrast agents
* pulmonary valve stenosis
* pulmonary embolism
* relevant tricuspid regurgitation
* cardiomyopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2006-06

CONTACTS AND LOCATIONS:
Overall Officials: Peter Schenk, MD, Principal Investigator — Intensive Care Unit 13h1, Dep. of Internal Medicine IV, Medical University of Vienna
Locations (1):
- Intensive Care Unit 13H1, Dep. of Internal Medicine IV, Medical University of Vienna, Vienna, Vienna, Austria

REFERENCES:
- [Background] Rodriguez-Roisin R, Krowka MJ, Herve P, Fallon MB; ERS Task Force Pulmonary-Hepatic Vascular Disorders (PHD) Scientific Committee. Pulmonary-Hepatic vascular Disorders (PHD). Eur Respir J. 2004 Nov;24(5):861-80. doi: 10.1183/09031936.04.00010904. No abstract available. PMID 15516683